CLINICAL TRIAL: NCT02425553
Title: Effects of Diet and Alcohol on Fullness, Reflux and Dyspeptic Symptoms After Meals
Brief Title: Effects of Diet on Reflux and Dyspepsia
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-Nr. 2015-0095
Record Dates: First submitted 2015-04-07; First posted 2015-04-24 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Gastroesophageal Reflux; Dyspepsia
Keywords: Diet; Reflux; Dyspepsia; Symptoms; Alcohol
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia | interventions — Diet; Meals

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Faculty and Delegates of Ascona II Meeting
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — High calorie (1200 kcal), high fat (50% energy), 400 ml juice (230 kcal)
  Other Names: Dinner
Other: Diet — High calorie (1200 kcal), low fat (20% energy), 400 ml juice (230 kcal)
  Other Names: Dinner
Other: Diet — Low calorie (600 kcal), low fat (20% energy), 400 ml juice (230 kcal)
  Other Names: Dinner
Other: Diet — High calorie (1200 kcal), high fat (50% energy), 300 ml wine (40 g alcohol, 230 kcal), 100 ml water
  Other Names: Dinner

SUMMARY:
Reflux and dyspeptic symptoms are common affecting 10-20% of the population on a regular basis. Reflux symptoms such as heartburn and regurgitation are caused by the return of acid or non-acid gastric contents into the esophagus. Dyspeptic symptoms are caused by abnormal gastric relaxation (impaired accommodation) or increased sensitivity of the stomach to distension during the meal.

The effects of diet on gastrointestinal function are debated and the efficacy of dietary management for digestive symptoms has not been established. Epidemiological studies suggest an effect; however, it is not possible to distinguish the effects of fat intake and total energy (i.e. calorie) intake in this work. This issue has been addressed by small physiological studies. The results show that esophageal acid exposure was related to total calorie intake but not to fat content. In contrast, the number of reflux symptoms was 40% higher after the high-fat than the low-fat meals. Similar findings were found for the relationship between gastric distension, fullness and dyspeptic symptoms by Magnetic Resonance Imaging. Thus, it appears that fat does not cause digestive dysmotility but heightens sensitivity to visceral events and so increases the number and severity of symptoms reported by patients. As yet, these findings have not been confirmed in larger, more representative surveys.

Similar to the effects of food, there are inconsistent findings regarding the effects of alcohol on gastro-esophageal reflux (GER) and gastric function. Physiological studies have noted delayed gastric emptying and an increase in reflux events when alcohol is taken with food. However, larger surveys have not confirmed that alcohol triggers reflux or dyspeptic symptoms.

The proposed observational, dietary study with cross-over design will assess the independent effects of energy intake (i.e. calorie load) and fat intake on gastric fullness, the number and severity of reflux and dyspeptic symptoms after meals. The effect of alcohol on symptoms after the high calorie, high fat meals will also be documented. The study population of senior academics attending a conference are likely to have a relatively high prevalence of risk factors for gastro-esophageal reflux disease (GERD) being predominantly male, with an older age and a larger waist circumference than average in the general community. This will increase study power and relevance of the findings.

The results will provide new information concerning the impact of dietary factors and alcohol on digestive symptoms after meals. This data will inform future guidelines for the dietary management of patients with reflux and dyspeptic symptoms after meals which will be relevant in both primary and secondary care.

DETAILED DESCRIPTION:
This is an observational, dietary study with cross-over design. Restaurant style meals and beverages are provided to faculty and delegates attending the Ascona II conference that agree to participate and provide written consent. Approximately 120 participants are expected to be recruited.

On four consecutive days the evening meal served will vary in calorie load and fat content using the established, partially balanced study design applied in previous studies. On the first three days fruit juice will be served, whereas, on the final day, an alcoholic beverage with the same acidity and number of calories will be served. All meals will have the same size and salt content. Controlling for all these parameters will reduce possible confounding factors in the analysis.

1. High calorie (1200 kcal), High fat (50% energy), 400 ml juice (230 kcal)
2. High calorie (1200 kcal), Low fat (20% energy), 400 ml juice (230 kcal)
3. Low calorie (600 kcal), Low fat (20% energy), 400 ml juice (230 kcal)
4. High calorie (1200 kcal), High fat (50% energy), 300 ml wine (40 g alcohol, 230 kcal), 100 ml water Note: The order of meals on day 1-3 will be fixed, but not necessarily in the order above. Meal constituents will not be disguised.

Note: Testing digestive symptoms in response to diet on successive days is possible because clinical physiological studies have shown no evidence of a sequence effect in previous studies using similar test meals.

An alginate-antacid preparation will be available as required for acute relief of any reflux or dyspeptic symptoms (Gaviscon Liquid, Reckitt Benckiser (available across-the-counter for this indication in Switzerland)). No participant is required to take this preparation.

The occurrence and severity of fullness, reflux and dyspeptic symptoms will be recorded contemporaneously by participants for three hours after each of the four test meals using a mobile application (SymTrack, Gastric Imaging & Analysis GmbH, Zürich, Switzerland). Paper forms will be made available for those without a mobile device. Three hours is the period of time during which reflux and dyspeptic symptoms are most often reported after meals. Positive reporting bias will be minimized by automatic reminders sent to the participants by the SymTrack every 30 minutes for three hours to remind participants to document the severity of symptoms including, if appropriate, an absence of symptoms. The use of the rescue medication to treat reflux and dyspeptic symptoms during the study will also be documented on the SymTrack. Symptoms and use of the rescue medication that occur after this three hour period up to 12 hours (i.e. the following morning) will be documented as part of safety follow-up data; however these will not contribute to primary or secondary outcomes.

All faculty and delegates will be invited to participate in this observational, dietary study. The investigators expect to recruit all, or nearly all, of those attending. The fixed menu provided every night by the restaurant will be the same whether the attendee does or does not participate in the study (unless specific dietary requirements are present). Involvement of almost all attendees will reduce selection bias; however, selection bias will remain because the group of clinical academics is not wholly representative of the general population. Note that the study population is predominantly male, with an older age and a larger waist circumference than the average in the community. These are all risk factors for reflux disease. This should increase study power to show treatment effect and the clinical relevance of findings.

All those attending the Centro Stefano Franscini conference centre in Ascona take their evening meal together. The cost of these meals is included in the registration package. This is a fixed menu with non-alcoholic drinks (alcohol is available to purchase). No other food is available on site except for individuals that have registered special dietary requirements. If other food is wanted, then this is available nearby in the town of Ascona. This local organizational arrangement with the provision of fixed meals free of charge will encourage compliance with the diet.

If the participants do not adhere to the meal and beverages set out in the study protocol then this can be documented using the SymTrack. To assess compliance, the participant will respond to the questions "did the patient consume the study meal?", "did the patient take additional food?", "did the patient consume the study beverage?", and "did the patient take additional alcoholic drinks?". Failure to comply with study procedures will not preclude the individual from participating on the following days.

The primary study analysis will investigate associations between number symptoms and caloric and fat content of the meals. It will be expressed as odds ratio. There will be a qualitative description of the deviation from study protocol. For example if participants report drinking alcohol during or after the meal on days 1-3 this will be expressed as a percentage deviation.

The primary and secondary variables plus other outcomes of interest will be documented using a mobile application (SymTrack; Gastric Imaging and Analysis GmbH, Zürich, Switzerland). Paper symptom diaries will be available for those participants without access to a smartphone.

On arrival at the meeting each attendee that agrees to participate and signs Written Informed Consent will be given personal instructions as to the operation of the mobile application. Should any difficulties remain then investigators, including those involved in the development of the app, will be on hand to assist participants.

Once the Written Informed Consent is signed the participants will be given a unique username and password to allow them to log into the SymTrack and start entering screening information and symptoms. This username will allow the identification of study participant as data is entered and ensure effective monitoring of data.

The primary analysis will be performed following study completion. The primary outcome is the number of reflux or dyspeptic symptoms. Odds ratio will be computed to describe the association of the number of symptoms with the meal calorie load and fat content.

Secondary outcomes are the severity of reflux and the severity of dyspeptic symptoms as well as sensation of fullness after each test meal. Analogue to the primary outcome an odds ratio will be computed to describe the association of these outcomes with the meal calorie load and fat content.

An odds ratio will be computed to describe the association of the primary and secondary outcomes with the ingestion of alcohol after the meal.

An additional analysis will be performed to identify factors - other than composition of the test meal - that increase the likelihood of reporting reflux and dyspeptic symptoms after meals (e.g. age, gender, BMI and low quality of life score).

Control questions that describe the study compliance will be described using descriptive statistics.

The majority of data acquired in this study originates from electronic sources. Screening data and symptoms entered via the smartphone are immediately transferred over an encrypted channel to the server and stored in a MySQL-database. Both the server application and the database are hosted on a professional application hosting provider located in Switzerland. The server application and the database design are developed and tested by Gastric Imaging & Analysis GmbH. The software version used during this study will be tested using semi-automated functional tests and load tests. Study principal investigator (Mark Fox) is responsible for all data stored in the database.

To ensure that the study is conducted in accordance with ethical principles, internal monitoring will be carried out regularly throughout the study. At the screening the internal monitor will review the protocol, and the database and all other aspects of the study with the investigator and other staff. Monitoring will be carried out early in the study and again after the last subject has completed the study. During monitoring, the monitor will verify compliance with the protocol and amendment(s), review the signed informed consent forms, diverse logs and all other source data. Direct access to all study-related site and source data/documents is mandatory for the monitoring review. Study team staff must be made available to answer any queries during the monitoring process.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be faculty and delegates attending the "Ascona II: Advances in clinical measurement of gastrointestinal motility and function" conference.

Exclusion Criteria:

* Age < 18,
* special dietary requirements incompatible with meals served at congress hotel restaurant,
* participation in another study with investigational drug within the 30 days preceding and during the present study (purely diagnostic studies are acceptable),
* individuals unwilling to provide written informed consent,
* inability to follow the procedures of the study, e.g. due to language problems (all study documents in English).

Participants with a history of alcohol dependency or medical conditions that may be exacerbated or affected by alcohol intake are allowed to participate but are instructed not to drink the alcohol provided with the high calorie, high fat test meal on day 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be all faculty and delegates attending the "Ascona II: Advances in clinical measurement of gastrointestinal motility and function" conference that agree to participate in the study and sign the informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of reflux symptoms | Participants will be followed for the duration of the conference, an expected average of 4 days
  Similar to "Pharmacokinetic outcome measures" the occurrence of reflux symptoms after each dinner will be summed up and compared between different dinners.
Number of dyspeptic symptoms | Participants will be followed for the duration of the conference, an expected average of 4 days
  Similar to "Pharmacokinetic outcome measures" the occurrence of dyspeptic symptoms after each dinner will be summed up and compared between different dinners.

SECONDARY OUTCOMES:
The severity of reflux symptoms measured by a visual-to-analogue scale from 0 to 100 | Participants will be followed at time points -30 min (before dinner) and at 0, 30, 60, 90, 120, 150, 180 min (after dinner) for 4 consecutive days
The severity of dyspeptic symptoms measured by a visual-to-analogue scale from 0 to 100 | Participants will be followed at time points -30 min (before dinner) and at 0, 30, 60, 90, 120, 150, 180 min (after dinner) for 4 consecutive days
The sensation of fullness measured by a visual-to-analogue scale from 0 to 100 | Participants will be followed at time points -30 min (before dinner) and at 0, 30, 60, 90, 120, 150, 180 min (after dinner) for 4 consecutive days

OTHER OUTCOMES:
Quality of Life measured by EQ-5D Quality of Life questionnaire | Participants will be followed for the duration of the conference, an expected average of 4 days
  A 5-item index score, the VAS score and the utility score (composite score calculated from the first two scores) from the EQ-5D Quality of Life questionnaire.
Postprandial Distress measured by Leuven dyspepsia questionnaire | Participants will be followed for the duration of the conference, an expected average of 4 days
  A composite score from Leuven dyspepsia questionnaire will be analysed
Safety outcome measured by the number of severe reflux symptoms | Participants will be followed for the duration of the conference, an expected average of 4 days
  Severe reflux symptom was defined as >60% on the visual-to-analogue scale form 0 to 100
Safety outcome measured by the number of severe dyspeptic symptoms | Participants will be followed for the duration of the conference, an expected average of 4 days
  Severe dyspeptic symptom was defined as >60% on the visual-to-analogue scale form 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Fox, Prof. (UK), Principal Investigator — Division of Gastroenterology and Hepatology, University Hospital Zurich, Switzerland

REFERENCES:
- [Background] Dent J, El-Serag HB, Wallander MA, Johansson S. Epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2005 May;54(5):710-7. doi: 10.1136/gut.2004.051821. PMID 15831922
- [Background] Fox M, Forgacs I. Gastro-oesophageal reflux disease. BMJ. 2006 Jan 14;332(7533):88-93. doi: 10.1136/bmj.332.7533.88. No abstract available. PMID 16410582
- [Background] DeVault KR, Castell DO; American College of Gastroenterology. Updated guidelines for the diagnosis and treatment of gastroesophageal reflux disease. Am J Gastroenterol. 2005 Jan;100(1):190-200. doi: 10.1111/j.1572-0241.2005.41217.x. PMID 15654800
- [Background] Tytgat GN, McColl K, Tack J, Holtmann G, Hunt RH, Malfertheiner P, Hungin AP, Batchelor HK. New algorithm for the treatment of gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2008 Feb 1;27(3):249-56. doi: 10.1111/j.1365-2036.2007.03565.x. Epub 2007 Oct 31. PMID 17973975
- [Background] Zheng Z, Nordenstedt H, Pedersen NL, Lagergren J, Ye W. Lifestyle factors and risk for symptomatic gastroesophageal reflux in monozygotic twins. Gastroenterology. 2007 Jan;132(1):87-95. doi: 10.1053/j.gastro.2006.11.019. Epub 2006 Nov 17. PMID 17241862
- [Background] Fox M, Barr C, Nolan S, Lomer M, Anggiansah A, Wong T. The effects of dietary fat and calorie density on esophageal acid exposure and reflux symptoms. Clin Gastroenterol Hepatol. 2007 Apr;5(4):439-44. doi: 10.1016/j.cgh.2006.12.013. Epub 2007 Mar 23. PMID 17363334